CLINICAL TRIAL: NCT01744704
Title: Phase I, Randomised, Double-masked, Placebo-controlled, Combined Single and Multiple Ascending Dose Study to Evaluate Safety, Tolerability and Pharmacokinetics of rhNGF Eye Drops in Healthy Male and Female Volunteers
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of rhNGF Eye Drops in Healthy Volunteers
Acronym: NGF0112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NGF0112; 2012-004302-10 (EudraCT Number)
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Nerve Growth Factor; Ophthalmic Solutions; Eye Drops; rh-NGF
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — cenegermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- rhNGF 0.5 µg/mL Sentinel (Experimental): 1 x 35 µL drop 3 subjects
  Interventions: Drug: rhNGF 0.5 µg/mL Sentinel
- rhNGF 5 µg/mL Sentinel (Experimental): 1 x 35 µL drop 3 subjects
  Interventions: Drug: rhNGF 5 µg/mL Sentinel
- rhNGF 60 µg/mL Part A (Experimental): 3 x 35 µL drops applied at 4 h intervals 6 subjects
  Interventions: Drug: rhNGF 60 µg/mL Part A
- rhNGF 20 µg/mL Sentinel (Experimental): 1 x 35 µL drop 3 subjects
  Interventions: Drug: rhNGF 20 µg/mL Sentinel
- rhNGF 20 µg/mL Part A (Experimental): 3 x 35 µL drops applied at 4 h intervals 6 subjects
  Interventions: Drug: rhNGF 20 µg/mL Part A
- rhNGF 180 µg/mL Part A (Experimental): 3 x 35 µL drops applied at 4 h intervals 6 subjects
  Interventions: Drug: rhNGF 180 µg/mL Part A
- Placebo Part A (Placebo Comparator): 3 x 35 µL drops applied at 4 h intervals 6 subjects
  Interventions: Drug: Placebo Part A
- rhNGF 20 µg/mL Part B (Experimental): 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 12 subjects
  Interventions: Drug: rhNGF 20 µg/mL Part B
- rhNGF 60 µg/mL Part B (Experimental): 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 9 subjects
  Interventions: Drug: rhNGF 60 µg/mL Part B
- rhNGF 180 µg/mL Part B (Experimental): 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 9 subjects
  Interventions: Drug: rhNGF 180 µg/mL Part B
- Placebo Part B (Placebo Comparator): 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 10 subjects
  Interventions: Drug: Placebo Part B

INTERVENTIONS:
Drug: rhNGF 0.5 µg/mL Sentinel — In Part 0, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration in the study eye (right or left) according to the randomisation list to achieve the required dose level
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 0.5 µg/mL Sentinel
Drug: rhNGF 5 µg/mL Sentinel — Part 0 represented a sentinel group.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 5 µg/mL Sentinel
Drug: rhNGF 20 µg/mL Sentinel — In Part 0, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration in the study eye (right or left) according to the randomisation list to achieve the required dose level
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 20 µg/mL Sentinel
Drug: rhNGF 20 µg/mL Part A — In Part A, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h on Day 1 to achieve the required fractionated single dose level.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 20 µg/mL Part A
Drug: rhNGF 60 µg/mL Part A — In Part A, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h on Day 1 to achieve the required fractionated single dose level.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 60 µg/mL Part A
Drug: rhNGF 180 µg/mL Part A — In Part A, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h on Day 1 to achieve the required fractionated single dose level.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 180 µg/mL Part A
Drug: rhNGF 20 µg/mL Part B — In Part B, as planned 3 dose levels of rh-NGF or placebo eye drops were studied in a total of 40 healthy subjects.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 20 µg/mL Part B
Drug: rhNGF 60 µg/mL Part B — In Part B, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h for 5 days to achieve the required multiple fractionated dose level.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 60 µg/mL Part B
Drug: rhNGF 180 µg/mL Part B — In Part B, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h for 5 days to achieve the required multiple fractionated dose level.
  Other Names: Recombinant Human Nerve Growth Factor
  Arms: rhNGF 180 µg/mL Part B
Drug: Placebo Part A — In Part A, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h on Day 1 to achieve the required fractionated single dose level.
  Other Names: Vehicle
  Arms: Placebo Part A
Drug: Placebo Part B — In Part B, all subjects received one 35-μL drop of rh-NGF at an appropriate concentration or placebo in their study eye (right or left) according to the randomisation list (and 1 drop of placebo in the non-study eye). This occurred q4h for 5 days to achieve the required multiple fractionated dose level.
  Other Names: Vehicle
  Arms: Placebo Part B

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of single and multiple ascending doses of rhNGF when administered as eye drops in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase I, randomised, double-masked, placebo-controlled eye drops administration study of rh-NGF in healthy male and female subjects.

This study consists of a single ascending dose part (part 0 one drop single application). Then single ascending dose part (part A; one drop three times a day) and a multiple ascending dose part (part B; one drop three times a day for five days). All parts of the study will consist of 3 ascending dose levels.

In order to support the dose escalation MAD phase from Covance, Basel to Covance, Leeds, an additional cohort (0M) will be conducted at Covance, Leeds at the same dose level as cohort 1M to ensure a degree of consistency between the two sites, i.e. that no dose escalation stopping criteria were met at either site.

In Part 0, each ascending dose cohort will include 3 subjects treated with one dose of rh-NGF.

In part A, each ascending dose cohort will include 6 subjects treated with rh-NGF and 2 with placebo.

In part B, each ascending dose cohort will include 9 subjects treated with rh-NGF drug and 3 with placebo, in addition to cohort 0M, which will include 3 subjects treated with rh-NGF and 1 with placebo

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 18 and 60 years, inclusive.
* Subject has to be able to communicate well with the investigator, understands and complies with the requirements of the study, and understands and signs the written volunteer informed consent form.
* Subject's systemic and ocular medical history must be considered normal in the opinion of the investigator at the Screening and Baseline visits.
* Best corrected distance visual acuity (BCDVA) score ≤ 0.00 LogMAR (≥83 ETDRS letters, 20/20 Snellen or 1.0 decimal fraction) in each eye at the Screening and Baseline visits.
* Normal anterior segment on external and slit lamp examination in both eyes at the Screening and Baseline visits.
* Normal posterior segment on fundus ophthalmoscopic examination in both eyes at the Screening and Baseline visits.
* Subject must be considered in good systemic health in the opinion of the investigator at the Screening and Baseline visits, as determined by:

  1. Subject's body mass index is between 18.5 and 30.4 kg/m2 inclusive
  2. A pre-study physical examination with no clinically significant abnormalities.
  3. Vital signs within clinically acceptable ranges for the purposes of the study (sitting systolic blood pressure [BP] ≥ 90 mmHg and ≤ 150 mmHg; diastolic BP ≥ 50 mmHg and ≤ 95 mmHg; heart rate (pulse rate) ≥ 40 and ≤ 100 beats per minute; oral body temperature ≥ 35.5°C and ≤ 37.5°C).
  4. An ECG with no clinically significant abnormalities, in the opinion of the Investigator.
  5. Pre-study clinical laboratory findings within normal range or not deemed clinically significant in the opinion of the investigator if outside of the normal range
* Female subjects will be:

  * either post menopausal where post menopause is defined as the period following peri-menopause, i.e. postmenopausal after 12 months without a menstrual period and with a serum FSH value within the reference range for postmenopausal females at Screening
  * or permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy)
  * or be using 2 different forms of highly effective contraception throughout the study.

Male subjects with female partners of child-bearing potential must use 2 different forms of highly effective contraception throughout the study and for a further 3 months after the follow-up visit and all male subjects must be willing to avoid donating sperm during this time.

Exclusion Criteria:

* Subject has had a clinically significant illness in the 6 weeks before screening in the opinion of the investigator.
* Subject is not suitable to participate in the study in the opinion of the investigator
* Subject has participated in any clinical study with an investigational drug/device within 3 months prior to the first day of dosing.
* Subject has had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or has a clinically significant allergy to drugs, foods or other materials (in the opinion of the investigator).
* Administration of any topical ocular (prescription or over the counter including artificial tears) or systemic medication including herbal product or fish oil preparations within 14 days before the first dose of study drug. Vitamins and mineral supplements not containing other substances are allowed until 96 hours before each dose if considered by the Investigator unlikely to interfere with the study results. Paracetamol at doses of at most 2 grams per day and ibuprofen at doses of at most 1200 mg per day for no more than 3 consecutive days or 6 non-consecutive days are allowed. Oral, injectable and implantable hormonal contraceptives are allowed without restrictions for female subjects. Longer exclusion periods apply for:

  1. amiodarone and hydroxychloroquine (210 days),
  2. monoclonal antibodies/ immunoglobulins/ other therapeutic proteins (120 days)
  3. Experimental drugs with a half life known to the Study Unit: Five half lives plus 2 weeks
  4. Experimental drugs with a half life unknown to the Study Unit: 120 days
  5. chloroquine and flunarizine (100 days)
  6. fluoxetine (75 days),
  7. benzodiazepines different from midazolam, lorazepam and triazolam, chlorpromazine, mephenytoin, nortryptyline, phenobarbital, primidone, carbamazepine, phenytoin and phenprocoumon (35 days).
* Subject has a significant history of drug/solvent abuse (within the last 2 years) or a positive drugs of abuse test at any time during the study.
* Subject has a history of alcohol abuse (within the last 2 years) or currently drinks in excess of 28 units per week or has a positive alcohol breath test at any time during the study.
* Subject is a smoker or has smoked in the 6 months prior to dosing.
* Subject who has a positive human immunodeficiency virus (HIV) screen, hepatitis B screen or hepatitis C screen.
* Subject has donated blood or blood products (e.g., plasma or platelets) within the 3 months prior to screening.
* Subject has a partner who will be pregnant or breastfeeding during the study
* Pregnant or breastfeeding female or those with a positive pregnancy test or who will not use a medically acceptable contraceptive method from selection and during the study
* Subject having used any glucocorticosteroid by any route in the last 30 days whichever the route of administration, or any medication by ocular or nasal administration route from 30 days before screening.
* Subjects currently diagnosed with any active ocular disease, even if mild, other than refractive error.
* Subject with history of ocular surgery, including laser refractive surgery
* Subject using a contact lens within 7 days prior administration of the first dose
* Intraocular pressure (IOP) >= 22 mmHg in either eye
* Presence of any corneal opacity or corneal fluorescein staining >0.5 grade using the modified Oxford scale
* Schirmer's test without anesthesia <= 9 mm/5 minutes
* Tear film break up time < 8 seconds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Kamtchoua, MD, Principal Investigator — Covance Basel Research Unit AG; Ashley Brooks, MBChB, Principal Investigator — Covance; Pier Adelchi Ruffini, MD, Study Director — Dompé s.p.a.Via San Martino, 12 - 20122 Milan, Italy; Mauro P Ferrari, PharmD, Study Director — Dompé s.p.a. - Via San Martino, 12 - 20122 Milan, Italy
Locations (2):
- Covance Basel Research Unit AG - Lettenweg 118 -, Allschwil, Switzerland
- COVANCE CLINICAL RESEARCH UNIT Ltd - Springfield House - Hyde Street, Leeds, United Kingdom

REFERENCES:
- [Background] Apfel SC, Kessler JA, Adornato BT, Litchy WJ, Sanders C, Rask CA. Recombinant human nerve growth factor in the treatment of diabetic polyneuropathy. NGF Study Group. Neurology. 1998 Sep;51(3):695-702. doi: 10.1212/wnl.51.3.695. PMID 9748012
- [Background] Apfel SC, Schwartz S, Adornato BT, Freeman R, Biton V, Rendell M, Vinik A, Giuliani M, Stevens JC, Barbano R, Dyck PJ. Efficacy and safety of recombinant human nerve growth factor in patients with diabetic polyneuropathy: A randomized controlled trial. rhNGF Clinical Investigator Group. JAMA. 2000 Nov 1;284(17):2215-21. doi: 10.1001/jama.284.17.2215. PMID 11056593
- [Background] Bonini S, Lambiase A, Rama P, Caprioglio G, Aloe L. Topical treatment with nerve growth factor for neurotrophic keratitis. Ophthalmology. 2000 Jul;107(7):1347-51; discussion 1351-2. doi: 10.1016/s0161-6420(00)00163-9. PMID 10889110
- [Background] Lambiase A, Rama P, Bonini S, Caprioglio G, Aloe L. Topical treatment with nerve growth factor for corneal neurotrophic ulcers. N Engl J Med. 1998 Apr 23;338(17):1174-80. doi: 10.1056/NEJM199804233381702. PMID 9554857
- [Background] Liu Q, McDermott AM, Miller WL. Elevated nerve growth factor in dry eye associated with established contact lens wear. Eye Contact Lens. 2009 Sep;35(5):232-7. doi: 10.1097/ICL.0b013e3181b3e87f. PMID 19672199
- [Background] Petty BG, Cornblath DR, Adornato BT, Chaudhry V, Flexner C, Wachsman M, Sinicropi D, Burton LE, Peroutka SJ. The effect of systemically administered recombinant human nerve growth factor in healthy human subjects. Ann Neurol. 1994 Aug;36(2):244-6. doi: 10.1002/ana.410360221. PMID 8053664
- [Background] Qi H, Li DQ, Shine HD, Chen Z, Yoon KC, Jones DB, Pflugfelder SC. Nerve growth factor and its receptor TrkA serve as potential markers for human corneal epithelial progenitor cells. Exp Eye Res. 2008 Jan;86(1):34-40. doi: 10.1016/j.exer.2007.09.003. Epub 2007 Sep 15. PMID 17980361
- [Background] Schifitto G, Yiannoutsos C, Simpson DM, Adornato BT, Singer EJ, Hollander H, Marra CM, Rubin M, Cohen BA, Tucker T, Koralnik IJ, Katzenstein D, Haidich B, Smith ME, Shriver S, Millar L, Clifford DB, McArthur JC; AIDS Clinical Trials Group Team 291. Long-term treatment with recombinant nerve growth factor for HIV-associated sensory neuropathy. Neurology. 2001 Oct 9;57(7):1313-6. doi: 10.1212/wnl.57.7.1313. PMID 11591856
- [Derived] Ferrari MP, Mantelli F, Sacchetti M, Antonangeli MI, Cattani F, D'Anniballe G, Sinigaglia F, Ruffini PA, Lambiase A. Safety and pharmacokinetics of escalating doses of human recombinant nerve growth factor eye drops in a double-masked, randomized clinical trial. BioDrugs. 2014 Jun;28(3):275-83. doi: 10.1007/s40259-013-0079-5. PMID 24327173

RESULTS

PARTICIPANT FLOW:
Groups:
- rhNGF 0.5 µg/mL Sentinel: 1 x 35 µL drop 3 subjects
  rhNGF 0.5 µg/mL Sentinel: one drop administration
- rhNGF 5 µg/mL Sentinel: 1 x 35 µL drop 3 subjects
  rhNGF 5 µg/mL Sentinel
- rhNGF 20 µg/mL Sentinel: 1 x 35 µL drop 3 subjects
  rhNGF 20 µg/mL Sentinel
- rhNGF 60 µg/mL Part A: 3 x 35 µL drops applied at 4 h intervals 6 subjects
  rhNGF 60 µg/mL Part A
- rhNGF 20 µg/mL Part A: 3 x 35 µL drops applied at 4 h intervals 6 subjects
  rhNGF 20 µg/mL Part A
- rhNGF 180 µg/mL Part A: 3 x 35 µL drops applied at 4 h intervals 6 subjects
  rhNGF 180 µg/mL Part A
- Placebo Part A: 3 x 35 µL drops applied at 4 h intervals 6 subjects
  Placebo Part A
- rhNGF 20 µg/mL Part B: 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 9 subject
  rhNGF 20 µg/mL Part B
- rhNGF 20 µg/mL Part B Cohort 0M: 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 3 subjects
  rhNGF 20 µg/mL Part B cohort 0M
- rhNGF 60 µg/mL Part B: 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 9 subjects
  rhNGF 60 µg/mL Part B
- rhNGF 180 µg/mL Part B: 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 9 subjects
  rhNGF 180 µg/mL Part B
- Placebo Part B: 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 10 subjects
  Placebo Part B
Period: Overall Study
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 60 µg/mL Part A | rhNGF 20 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 20 µg/mL Part B Cohort 0M | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Started | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 9 | 3 | 9 | 9 | 10
Completed | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 9 | 3 | 9 | 9 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | rhNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7) | 47 (9.2) | 29 (11.9) | 46 (10) | 36 (9.4) | 42 (17.8) | 42 (9) | 41 (12.1) | 36 (14.7) | 29 (10.3) | 36 (12.6) | 40.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 1 | 3 | 2 | 4 | 5 | 1 | 2 | 24
  Male | 1 | 1 | 2 | 5 | 5 | 4 | 4 | 8 | 4 | 8 | 8 | 50
Region of Enrollment [Number; unit: participants]
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 9 | 8 | 29
  Switzerland | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 9 | 0 | 0 | 2 | 45

OUTCOME MEASURES:

1. Primary Outcome: Changes in VAS Ocular Tolerability
Description: A global ocular discomfort score was determined using a 100 mm visual analogue scale (VAS) on which 0 means no symptoms and 100 means the worst possible discomfort. This evaluation was performed before any ophthalmic assessment at a given study visit. Specific ocular symptoms to be assessed with the VAS included: foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, photophobia.
  Part 0: VAS evaluated on days -1, 1, 3, 10 (FU) Part A: VAS evaluated on days -1, 1, 3, 10 (FU) Part B: VAS evaluated on days -1, 1, 5, 15 (FU) Follow up (FU) refers to participants' last available assessment.
  The Outcome Measure Time Points and Data Table refers to Part B.
Time Frame: Day -1, Day 1, Day 5, Day 15 (FU)
Population: Safety population: consisted of all subjects randomised into the study and receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | rhNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10
units on a scale
  Foreign body sensation - Day 1 (8h) vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 3 (7.3) | 0 (0) | 0 (0) | 0.4 (0) | 0 (0) | 0 (0.5) | 0 (0.5) | 0 (0.8)
  Foreign body sensation - Day 5 vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2.6) | 0 (0.5) | 0 (0.7) | 0 (0.7)
  Foreign body sensation - FU vs Day -1 | -1 (1.2) | 0 (0) | 0 (0.6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.5) | 0 (0.4) | 0 (0.6)
  Burning/Stinging - Day 1 (8h) vs Day -1 | -1 (1.2) | 0 (0) | 0 (0.6) | 2 (4.9) | 0 (0) | 0 (0) | 0 (0) | 0 (0.3) | 0 (0.5) | 0 (0.6) | 0 (0.3)
  Burning/Stinging - Day 5 vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3.5) | 0 (0.4) | 0 (0.5) | 0 (0.4)
  Burning/Stinging - FU vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.3) | 0 (0.5) | 0 (0.4) | 0 (0.6)
  Itching - Day 1 (8h) vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0.3) | 0 (0.3) | 0 (0.7) | 0 (0.4)
  Itching - Day 5 vs Day -1 | -1 (1.2) | 0 (0) | 0 (0.6) | 0 (0) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0.3) | 0 (0.3) | 0 (0.4) | 0 (0.5)
  Itching - FU vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.3) | 0 (0.7) | 0 (0.6) | 0 (0)
  Pain - Day 1 (8h) vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0.3) | 0 (0.7) | 0 (0.7) | 0 (0.8)
  Pain - Day 5 vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0.3) | 1 (3.5) | 4 (6.5) | 0 (1.1)
  Pain - FU vs Day -1 | -1 (1.2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0.3) | 0 (0.7) | 0 (0.4) | 0 (0.7)
  Sticky feeling - Day 1 (8h) vs Day -1 | -1 (1.7) | 0 (0) | -3 (4.6) | -1 (1.6) | 0 (0.8) | 0 (0) | 1 (2.4) | 0 (0) | 0 (0.7) | 3 (7.6) | 0 (0.4)
  Sticky feeling - Day 5 vs Day -1 | -1 (1.7) | 0 (0) | -2 (4.9) | -1 (1.6) | 0 (0.8) | 0 (0) | 0 (0.4) | 0 (0.3) | 0 (0.5) | 1 (3.6) | 0 (0.6)
  Sticky feeling - FU vs Day -1 | -1 (1.7) | 0 (0) | -3 (4.6) | -1 (1.6) | 0 (0.8) | 0 (0) | 0 (0.4) | 0 (0.3) | 0 (0.5) | 0 (0.4) | 0 (0.3)
  Blurred vision - Day 1 (8h) vs Day -1 | -2 (1.5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0) | 0 (0.5) | 0 (0.3) | 0 (0.5)
  Blurred vision - Day 5 vs Day -1 | -2 (1.5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0.3) | 0 (0.5)
  Blurred vision - FU vs Day -1 | -2 (1.5) | 0 (0) | 0 (0.6) | 0 (0.4) | 0 (0) | 0 (0) | 0 (0.4) | 0 (0) | 0 (0.3) | 1 (0.5) | 0 (0.5)
  Photophobia - Day 1 (8h) vs Day -1 | -1 (1.7) | 0 (0) | 0 (0) | 1 (3.3) | 1 (1.6) | 0 (0) | 0 (0) | 0 (0) | 0 (0.5) | 0 (0.6) | 0 (0.5)
  Photophobia - Day 5 vs Day -1 | -1 (1.7) | 0 (0) | 0 (0.6) | 0 (0) | 0 (0) | 0 (0) | 0 (0.8) | 1 (2.0) | 0 (0.5) | 0 (0.7) | 0 (0.5)
  Photophobia - FU vs Day -1 | -1 (1.7) | 0 (0) | 0 (0) | 0 (0) | 0 (0.8) | 0 (0) | 0 (0.4) | 0 (0) | 0 (0.7) | 0 (0.7) | 0 (0.5)

2. Primary Outcome: Change in Best Corrected Distance Visual Acuity (BCDVA)
Description: Best corrected distance visual acuity measured using the ETDRS (Early Treatment Diabetic Retinopathy Study) score. In this population, the scores range from -6 (worse visus) to 3 (best visus).
  The study includes Part 0, Part A and Part B. In Part B BCDVA was evaluated on days -1, 1, 5, 15 (FU). Follow up (FU) refers to participants' last available assessment.
Time Frame: Day -1, Day 1, Day 5, Day 15 (FU)
Population: Safety population consisted of all subjects randomised into the study and receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | rhNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10
units on a scale
  Day 1 vs Day-1 | 1 (0.6) | 3 (0.6) | -6 (3.1) | 3 (1.6) | 0 (0.4) | -0 (1.4) | 1 (1.6) | 1 (2.7) | 0 (3.7) | 0 (3.6) | 0 (3.1)
  Day 5 vs Day-1 | 1 (2.3) | 0.0 (4.7) | 1 (2.1) | 1 (2.6) | 1 (2.5) | 0 (2.8) | -1 (2.0) | 1 (2.7) | 1 (2.9) | 0 (3.3) | 0 (3.8)
  Day 15 (FU) vs Day-1 | 2 (2.5) | 2 (1.0) | -1 (2.9) | 2 (4.0) | 2 (1.9) | 0 (2.3) | 0 (3.2) | 1 (2.4) | 1 (2.4) | 2 (3.7) | 0 (2.1)

3. Primary Outcome: Change in Mean Tear Film Break up Time (TFBUT)
Description: Tear film break-up time was assessed by slit lamp examination (SLE). The shorter is the tear film break-up time, the worse is the dry eye symptom severity.
  The study includes Part 0, Part A and Part B. In Part B this endpoint was evaluated on days -1, 1, 5, 15 (FU). Follow up (FU) refers to participants' last available assessment.
Time Frame: Day -1, Day 1, Day 5, Day 15 (FU)
Population: Safety population: consisted of all subjects randomised into the study and receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | rhNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10
seconds
  Day 1 vs Day -1 | 1.7 (1.89) | 0.0 (0.5) | -2.6 (2.95) | 0.4 (0.86) | -0.5 (0.64) | -0.4 (1.93) | 0.0 (0.67) | 0.5 (1.14) | 0.4 (0.96) | 0.1 (1.11) | 0.2 (0.79)
  Day 5 vs Day -1 | -1.2 (1.62) | -0.3 (1.04) | 0.9 (1.21) | 0.1 (0.69) | -0.1 (0.85) | 0.0 (1.64) | -0.7 (1.53) | -0.2 (1.76) | -0.4 (1.52) | 0.2 (2.03) | -0.2 (1.03)
  Day 15 (FU) vs Day -1 | -1.4 (1.65) | 0.2 (0.29) | -0.9 (1.4) | -0.1 (1.32) | 0.4 (0.77) | -0.6 (0.69) | 1.0 (1.22) | 0.1 (1.07) | -0.4 (1.83) | -0 (1.48) | 0.0 (1.08)

4. Primary Outcome: Change in Mean Corneal Fluorescein Staining
Description: Slit lamp examination was used to assess the eyelid margin, conjunctiva, cornea, anterior chamber, iris and lens with the instillation of fluorescein to evaluate corneal fluorescein staining (modified Oxford scale).
  This is 7-point ordinal scale that scores 0, 0.5, and 1 to 5. On this scale the score 0 corresponds to no staining dots (complete corneal clearing) and the score 0.5 corresponds to three or less staining dots. The higher is the number of dots, the higher and worse is the score.
  The study includes Part 0, Part A and Part B. In Part B the endpoint was evaluated on days -1, 1, 5, 15 (FU).
Time Frame: Day -1, Day 1, Day 5, Day 15 (FU)
Population: Safety population: consisted of all subjects randomised into the study and receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- hNGF 60 µg/mL Part A: 3 x 35 µL drops applied at 4 h intervals 6 subjects rhNGF 60 µg/mL Part A
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | hNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10
Units on a scale
  Day 1 vs Day -1 | 1.7 (1.89) | 0.0 (0.50) | -2.6 (2.95) | 0.4 (0.86) | -0.5 (0.64) | -0.4 (1.93) | 0.0 (0.67) | 0.2 (1.14) | 0.4 (0.96) | 0.1 (1.11) | 0.2 (0.79)
  Day 5 vs Day -1 | -1.2 (1.62) | -0.3 (1.04) | -0.9 (1.21) | 0.1 (0.69) | -0.1 (0.85) | 0.0 (1.64) | -0.7 (1.53) | -0.2 (1.76) | -0.4 (1.52) | -0.2 (2.03) | -0.2 (1.03)
  Day 15 (FU) vs Day -1 | -1.4 (1.65) | 0.2 (0.29) | -0.9 (1.40) | -0.1 (1.32) | 0.4 (0.77) | -0.6 (0.69) | 1.0 (1.22) | 0.1 (1.07) | -0.4 (1.83) | -0.0 (1.48) | 0.0 (1.08)

5. Primary Outcome: Change in Intraocular Pressure (IOP)
Description: Intraocular pressure was determined using Goldmann applanation tonometry. The study includes Part 0, Part A and Part B. In Part B this endpoint was evaluated at screening and on days 7, 15 (FU).
  Follow up (FU) refers to participants' last available assessment.
Time Frame: Screening, Day 7, Day 15 (FU)
Population: Safety population: consisted of all subjects randomised into the study and receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | rhNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10
mmHg
  Day 7 vs screening | 1 (2.0) | -1 (1.5) | -1 (2.6) | 1 (1.8) | 1 (3.9) | 1 (1.6) | -2 (1.8) | -1 (2.0) | 0 (3) | -2 (3.7) | -2 (2.8)
  Day 15 (FU) vs screening | -1 (2.5) | 1 (0.6) | -1 (1.0) | 1 (2.7) | -1 (3.3) | 1 (3.2) | -2 (2.8) | 0 (5.3) | -1 (3.3) | -1 (3.1) | -3 (3.4)

6. Primary Outcome: Percentage of Abnormal Findings in Dilated Fundus Ophthalmoscopy
Description: Dilated fundus ophthalmoscopy (DFO) is used to view the eye's interior, allowing assessment of the retina/macula/choroid, optic nerve head, blood vessels, and other features.
  The outcome can be normal or abnormal. The study includes Part 0, Part A and Part B. In Part B this endpoint was evaluated on day 7.
Time Frame: Part B - Day 7
Population: Safety population: consisted of all subjects randomised into the study and receiving a dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage of abnormal findings
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 60 µg/mL Part A | rhNGF 20 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 12 | 9 | 9 | 10
percentage of abnormal findings | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Groups:
- rhNGF 20 µg/mL Part B: 3 x 35 µL drops applied at 4 h intervals per day during 5 consecutive days 12 subject
  rhNGF 20 µg/mL Part B
Arm/Group | rhNGF 0.5 µg/mL Sentinel | rhNGF 5 µg/mL Sentinel | rhNGF 20 µg/mL Sentinel | rhNGF 20 µg/mL Part A | rhNGF 60 µg/mL Part A | rhNGF 180 µg/mL Part A | Placebo Part A | rhNGF 20 µg/mL Part B | rhNGF 60 µg/mL Part B | rhNGF 180 µg/mL Part B | Placebo Part B
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/7 | 0/6 | 0/12 | 0/9 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 1/6 | 0/6 | 2/7 | 3/6 | 8/12 | 6/9 | 7/9 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | rhNGF 0.5 µg/mL Sentinel (N=3) | rhNGF 5 µg/mL Sentinel (N=3) | rhNGF 20 µg/mL Sentinel (N=3) | rhNGF 20 µg/mL Part A (N=6) | rhNGF 60 µg/mL Part A (N=6) | rhNGF 180 µg/mL Part A (N=7) | Placebo Part A (N=6) | rhNGF 20 µg/mL Part B (N=12) | rhNGF 60 µg/mL Part B (N=9) | rhNGF 180 µg/mL Part B (N=9) | Placebo Part B (N=10)
Abnormals sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1/6 (1) | 0/7 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal staining (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orapharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
No limitations and caveats area defined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No